CLINICAL TRIAL: NCT02564185
Title: Prospective, Randomized Study of the Impact of a Education Program for Patients Suffering From Low Back Pain
Acronym: TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/51; 2009-A01193-54 (Other: ANSM)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): The "control" group will follow usual practice.
  Interventions: Other: Usual practice
- Education program (Experimental): The "Education program" group benefit in addition of a therapeutic education program including nursing follow-up at 1, 3 and 6 months.
  Interventions: Other: Usual practice; Other: Education program

INTERVENTIONS:
Other: Usual practice
Other: Education program
  Arms: Education program

SUMMARY:
According to the WHO, therapeutic education is intended to help patients acquire or maintain the skills they need to optimally manage living with a chronic disease. Low back pain is frequent and therapeutic education could be a promising option.

The purpose of the study is to evaluate the impact of a therapeutic education program for patients suffering from low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain
* Treatment with transcutaneous electrical nerve stimulation (TENS)

Exclusion Criteria:

* Contra-indication of TENS
* Patients with mental disorders
* Lack of autonomy or patients living alone at home without help
* Concomitant inclusion in another research on the treatment of pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | 6 months
  EIFEL functional disability scale (Gagnon et al, Annals Phys Med Rehab, 2009, 1, 3-16).
Quality of life | 6 months
  DRAD questionnaire (Lawlis et al, Spine 1989;14:511-6.)

SECONDARY OUTCOMES:
Pain | 6 months
  Numerical scale
Neuropathic pain | 6 months
  DN4 questionnaire
Social impact | 6 months
  Changes in the employment status
Evaluation of the program | 6 months
  Self-administered questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France